CLINICAL TRIAL: NCT03517033
Title: An Open Label, Randomized, 2 -Period, 2 -Treatment, 2- Sequence, Crossover, Single-Dose BE Study of Nebivolol 20 mg Tablet [Torrent, India] Vs Bystolic® 20 mg Tablet [ Forest Pharmaceuticals Inc., USA] in Healthy Subjects Fed Condition.
Brief Title: Bioequivalence Study of Torrent Pharmaceuticals Ltd's Nebivolol 20 mg Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK-12-151
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Torrent's Nebivolol Tablets 20 mg
  Interventions: Drug: Torrent's Nebivolol Tablets
- Reference (Active Comparator): Forest Pharmaceuticals Inc's Bystolic Tablets 20 mg
  Interventions: Drug: Forest Pharmaceuticals Inc.'s Bystolic Tablets

INTERVENTIONS:
Drug: Torrent's Nebivolol Tablets
  Arms: Test
Drug: Forest Pharmaceuticals Inc.'s Bystolic Tablets
  Arms: Reference

SUMMARY:
Subjects to compare the single dose bioavailability of Torrent's Nebivolol Tablets 20 mg and Bystolic®20 mg Tablets of Forest Pharmaceuticals Inc., USA. Dosing periods of studies were separated by a washout period of 11 days.

DETAILED DESCRIPTION:
An Open Label, Randomized, 2- Period, 2 -Treatment, 2 -Sequence, Crossover, Single- dose Bioequivalence study of Nebivolol Tablets containing Nebivolol 20 mg (Test Formulation, Torrent Pharmaceuticals Ltd., India) Versus Bystolic® 20 mg Tablets containing Nebivolol 20 mg (Reference, Forest Pharmaceuticals Ltd., USA) in Healthy Volunteers Under Fed Condition.

ELIGIBILITY:
Inclusion Criteria:

* Sex: male
* Age: 18-45 years (inclusive both)
* Volunteer with BMI of 18-27 (inclusive both) kg/m2 with minimum of 50 kg weight.
* Healthy and willing to participate in the study.
* Volunteer willing to adhere to the protocol requirements and to provide written informed consent.
* Non-smokers or smoker who smokes less than 10 cigarettes per day.

Exclusion Criteria:

* Inability to communicate or co-operate.
* Volunteers suffering from any chronic illness such as arthritis, asthma etc.
* History of pre-existing bleeding disorder.
* Clinically relevant abnormalities in the results of the laboratory screening evaluation.
* Clinically significant abnormal ECG or Chest X-ray.
* HIV, HCV, HBsAg positive volunteers.
* History of significant blood loss due to any reason, including blood donation in the past 3 months.
* Participation in any study within past 3 months before entry to the study,
* History of alcohol or drug abuse.
* History of consumption of prescribed medication since last 14days or OTC medication/ herbal remedies since last 7 days before beginning of the study.
* Positive to breath alcohol test.
* Volunteer found to be positive for Opiate, tetra hydrocannabinol, amphetamine, barbiturates, benzodiazepines, Cocaine positive volunteers based on urine test.
* Systolic blood pressure less than 100 mmHg or more than 140 mmHg and diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
* Pulse rate less than 50/minute or more than 100/minute.
* Oral temperature less than 95°F or more than 98.6°F.
* Respiratory rate less than 12/minute or more than 20/minute.
* History of allergy to the test drug or any drug chemically similar to the drug under investigation.
* Recent History of kidney or liver dysfunction.
* Volunteers suffering from any psychiatric (acute or chronic) disorder.
* Existence of any surgical or medical condition, which, in the judgment of the Chief Investigator and/or clinical investigator/physician, might interfere with the absorption; distribution,· metabolism or excretion of the drug or likely to compromise the safety of Volunteers.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose to 72 hours post-dose
AUC | pre-dose to 72 hours post-dose